CLINICAL TRIAL: NCT05966792
Title: The Clinical Efficacy and Mechanism of SGLT2 Inhibitors Treating Polycystic Ovary Syndrome by Modulating the Nod-like Receptor Protein 3 Inflammasome
Brief Title: SGLT2 Inhibitors in Treating Patients With PCOS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Director, principal investigator, clinical professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGLT2i in PCOS
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Sodium-Glucose Transporter 2 Inhibitors; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGLT2 inhibitors (Experimental): Intervention with henggliflozin (10mg qd) for 6 months
  Interventions: Drug: SGLT2 inhibitors
- metformin (Placebo Comparator): Intervention with metformin (500mg bid) for 6 months
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: SGLT2 inhibitors — Sodium-glucose cotransporters inhibitors (SGLT2i) are novel hypoglycemic drugs with unique hypoglycemic mechanisms, which are completely independent of islet β-cell function or insulin sensitivity. Previous studies have shown that SGLT2i may improve IR by inhibiting glucotoxicity, reducing body weight, reducing inflammation, improving islet β-cell function, and reducing oxidative stress.
  Arms: SGLT2 inhibitors
Drug: metformin — Metformin is a classic drug for the treatment of polycystic ovary syndrome, which can improve the degree of insulin resistance in PCOS patients.
  Arms: metformin

SUMMARY:
Chronic inflammation is the core of Polycystic ovary syndrome (PCOS), and obesity and overweight further exacerbate the level of inflammation in the peripheral circulation and ovarian tissue in PCOS patients. Metformin is a classic endocrine drug for the treatment of PCOS, but its clinical response rate is only about 40%. Our previous published study (Diabetes Obes Metab, 2022) observed that the new hypoglycemic drug SGLT-2 inhibitor can significantly improve the clinical symptoms of patients with insulin resistance PCOS, and the clinical efficacy is not inferior to metformin, but its specific mechanism of action is not clear. Recent studies have shown that SGLT-2 significantly attenuates the activation of the Nod-like receptor protein 3 (NLRP3) inflammasomes and the secretion of IL-1β in patients with type 2 diabetes mellitus at high risk of cardiovascular disease. Based on the above research background, this project will combine clinical research and mechanism exploration to solve the following two problems:

1. whether SGLT2 inhibitor can further improve the clinical efficacy of PCOS patients compared to metformin;
2. mechanistic studies further clarify whether SGLT2 inhibitors improve inflammatory symptoms by modulating NLRP3 inflammosomes in the treatment of polycystic ovary syndrome;

DETAILED DESCRIPTION:
This clinical study is a prospective, single-center, randomized (1:1) controlled clinical study. The enrollment population is overweight or obese PCOS patients. After signing the informed consent form, patients who meet the inclusion/exclusion criteria will be randomly assigned to the experimental and control groups for treatment in a 1:1 ratio, for a total of 108 patients enrolled.

Subjects randomized to the trial group will receive SGLT-2 inhibitors for 24 weeks.

Participants randomised to control will receive metformin for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-45
* Meet Rotterdam criteria
* BMI≥20kg/m2

Exclusion Criteria:

* Treatment with any additional medications that might impede the trial, including GLP-1 RAs, metformin, pioglitazone, contraceptives, or traditional Chinese medicine within the past 3 months
* Pregnancy or lactation
* Mental illness
* Malignant tumors
* Chronic kidney disease or severe liver dysfunction
* Inflammatory bowel disease
* Involvement in other research programs within the past 3 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Menstrual cycles | 6 months
  annual number of menstrual cycles

SECONDARY OUTCOMES:
HOMA-IR | 6 months
  Homeostatic model assessment insulin resistance index
NLRP3 | 6 months
  serum Nod-like receptor protein 3
IL-1β | 6 months
  serum Interleukin-1 beta
IL-18 | 6 months
  serum Interleukin-18
LH | 6 months
  luteinizing hormone
FSH | 6 months
  follicle-stimulating hormone
PRL | 6 months
  prolactin
E2 | 6 months
  estradiol
P | 6 months
  progesterone
TT | 6 months
  total testosterone
AMH | 6 months
  antimullerian hormone antimullerian hormone antimullerian hormone antimullerian hormone

CONTACTS AND LOCATIONS:
Overall Officials: Manna Zhang, PhD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People'S Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No